CLINICAL TRIAL: NCT00681382
Title: INSPIRE Asthma Patient Survey to Clarify the Use of Asthma Medication and Effects of Asthma in Everyday Life in Finland
Brief Title: Asthma Patient Survey Study to Assess Asthma Effect and Medication in Finland
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Klaus Tamminen - MC Medical Director, AstraZeneca
Other Study IDs: NIS-RFI-SYM-2006/1
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma; use of asthma medication; asthma control; telephone survey; patient's perception
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Asthma patients using inhaled steroids as maintenance treatment

SUMMARY:
This study was aimed at clarifying how the asthma medication is used in practice and how asthma affects everyday life. Total of 106 GPs were asked to recruit patients using inhaled steroid as maintenance treatment for asthma to take part in a telephone survey. Altogether 142 patients were interviewed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed persistent asthma
* regular use of inhaled steroids and concomitant medication

Exclusion Criteria:

* never been diagnosed COPD
* seasonal asthma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Patients perceptions about treatment of asthma, asthma medication and what are the most common triggers that cause exacerbations. | Single occasion

SECONDARY OUTCOMES:
How patients react to the first signs of worsening of asthma i.e. how they use asthma medication during stable phase and asthma exacerbation | Single occasion
How asthma affects everyday life | Single occasion

CONTACTS AND LOCATIONS:
Overall Officials: Airi Puhakka, Study Director — AstraZeneca Finland; Jouni Hedman, Principal Investigator — South Karelia Central Hospital, Finland